CLINICAL TRIAL: NCT05738668
Title: Clinical-immunological Features of Anti-NMDAR Encephalitis
Acronym: Bio-NMDAr
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 750
Record Dates: First submitted 2022-09-05; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-09

CONDITIONS: Anti NMDA Receptor Encephalitis
Keywords: Anti NMDA Receptor Encephalitis; antibodies; relapses; outcomes
MeSH Terms: conditions — Anti-N-Methyl-D-Aspartate Receptor Encephalitis; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood, DNA, cells, CSF collected at diagnosis time
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anti-NMDAR encephalitis: Patients with well-characterized anti-NMDAR encephalitis.
  Interventions: Other: Description of clinical characteristic

INTERVENTIONS:
Other: Description of clinical characteristic — This is a non-interventional study involving clinical data and biological samples (blood, DNA, CSF). Clinical data are collected for the center and samples are already stored in biobank repositories and collected as part of "good clinical practice" in the diagnostic process of patients with suspected autoimmune encephalitis, meaning that the standard diagnostic and therapeutic approaches will not be altered in the selected study population. Patients have already gave explicit written consent for biological specimens sampling and storage at the "Centre de Ressources Biologiques des Hospices Civils de Lyon" (CRB-HCL) (including tissue, cells or biological fluids) and genetic analysis for research purposes. Additionally, patients will be informed about the present study.

SUMMARY:
Using a retrospective cohort of 501 patients with anti-NMDAR encephalitis to assess clinical and immunological prognostic biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Patient with neurological disorder
* Patient with NMDAR antibodies in sera or CSF

Exclusion Criteria:

* - No available clinical data
* Patient without NMDAR antibodies or neurological disorder

Age Groups: Child, Adult, Older Adult
Study Population: Patients with well-characterized anti-NMDAR encephalitis
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin scale (mRS) | Baseline
  Scale for measuring the degree of dependence in the daily activities of people who have suffered of neurological disability.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Neurologique Pierre Wertheimer / Groupement Hospitalier Est, Lyon, BRON, France